CLINICAL TRIAL: NCT06018012
Title: Magnetic Resonance Spectroscopy and Auditory Brain- Stem Response Audiometry as Early Predictors of Bilirubin-Induced Neurologic Dysfunction in Full-term Jaundiced Neonates
Brief Title: MRA and ABR as Early Predictors of Bilirubin-Induced Neurologic Dysfunction in Full-term Jaundiced Neonates
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Lamiaa Khaled Zidan, Assistant lecturer, Tanta University
Other Study IDs: MRS& ABR in jaundiced neonates
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1 or acute bilirubin encephalopathy: Group (1): included 26 cases with BIND or acute bilirubin encephalopathy (ABE).
  Interventions: Device: MRS and ABR
- 2 or neonatal hyperbilirubinemia: Group (2): included 30 cases with neonatal hyperbilirubinemia on
  Interventions: Device: MRS and ABR
- Control: control group: 20 healthy, age-matched neonates
  Interventions: Device: MRS and ABR

INTERVENTIONS:
Device: MRS and ABR — Magnetic Resonance Spectroscopy and Auditory Brain- stem Response Audiometry

SUMMARY:
The aim of the research was to define the role of MRS and ABR as early predictors of bilirubin-induced neurologic dysfunction (BIND) in full-term neonates who required intervention (phototherapy or exchange transfusion).

DETAILED DESCRIPTION:
Neonatal jaundice is a prevalent condition. It's typically a harmless phase that occurs as the body adjusts to bilirubin levels after birth, representing a balance between its production and elimination. When there's an increase in bilirubin production and a decrease in elimination, infants become at risk for dangerous hyperbilirubinemia, potentially leading to bilirubin encephalopathy.

The range of neurological issues caused by excessive bilirubin is referred to as bilirubin-induced neurologic dysfunction. Detecting this condition early is crucial to prevent irreversible brain damage. Some of the neurological effects include gliosis, demyelination, and interference with glutamate uptake by astrocytes in the basal ganglia. Magnetic resonance spectroscopy (MRS) is an advanced imaging technique that holds promise for identifying these metabolic changes and aiding in the diagnosis and evaluation of neonates with hyperbilirubinemia.

Bilirubin neurotoxicity particularly affects the auditory system, starting with the brainstem cochlear nuclei, followed by the auditory nerve. This damage can occur even without the classic signs of bilirubin encephalopathy and is known as auditory neuropathy spectrum disorder (ANSD). ANSD is characterized by abnormal auditory neural function, while cochlear microphonics and otoacoustic emissions remain normal.

The impact on hearing can vary from subtle issues in sound processing to complete deafness. Abnormal results in auditory brainstem response (ABR) tests can indicate the presence of acute bilirubin encephalopathy (ABE), serving as the most common and earliest sign of ABE.

ELIGIBILITY:
Inclusion Criteria:

* This study included term, appropriate for gestational age (AGA) neonates with pathological unconjugated hyperbilirubinemia who were candidates for intervention (Intensive phototherapy versus Exchange transfusion) using the American Academy of Pediatrics guidelines; 2004.

Exclusion Criteria:

1. Preterm neonates (less than 37 weeks).
2. Clinically moderate and severe acute bilirubin encephalopathy according to modified Bilirubin-induced neurologic dysfunction (BIND-M) score.
3. Neonates born with birth asphyxia and/or poor Apgar score.
4. Neonates with sepsis including CNS infection.
5. Neonates with family history of childhood hearing loss.
6. Congenital infection.
7. Chromosomal abnormalities.
8. Congenital ear anomalies associated with hearing loss or brain abnormalities including craniofacial anomalies.
9. Patients who were receiving ototoxic drugs as aminoglycosides.
10. Conjugated hyperbilirubinemia.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study included term, appropriate for gestational age (AGA) neonates with pathological unconjugated hyperbilirubinemia who were candidates for intervention (Intensive phototherapy versus Exchange transfusion) using the American Academy of Pediatrics guidelines; 2004. In addition, 20 healthy, age-matched neonates were included as controls.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Early detection of neurological abnormalities using MRS metabolic ratios in high-risk neonates without oblivious clinical signs | 2 years
  Early detection of neurological abnormalities in high-risk neonates, without oblivious clinical signs, chemically by using MRS metabolic ratio ( low NAA/Cr, NAA/Cho ratios, and high Lac/Cr ratio).
Early detection of neurological abnormalities using ABR parameters in high-risk neonates without oblivious clinical signs | 2 years
  Early detection of neurological abnormalities in high-risk neonates, without oblivious clinical signs, functionally through ABR parameters ( prolonged wave III peak latency, wave V peak latency, I-III interpeak interval, and I-V interpeak interval )
Bilirubin level and auditory abnormality | 2 years
  Finding out the lowest level of total serum bilirubin at which auditory pathway abnormality was found, in comparison to age.
Bilirubin level and MRS abnormality | 2 years
  Finding out the lowest level of total serum bilirubin at which MRS abnormalities were found, in comparison to age.

SECONDARY OUTCOMES:
Discriminative capacity of MRS for acute bilirubin encephalopathy | 2 years
  Determining the discriminative capacity of MRS metabolic ratios (NAA/Cr and NAA/Cho) for neonates with acute bilirubin encephalopathy and those without it with identification of the cutoff value those ratios at which acute bilirubin encephalopathy is present.
Discriminative capacity of ABR for acute bilirubin encephalopathy | 2 years
  Determining the discriminative capacity of ABR wave latencies and interpeak intervals abnormalities for neonates with acute bilirubin encephalopathy and those without it with identification of the cutoff value those latencies and intervals at which acute bilirubin encephalopathy is present.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine,Tanta University, Tanta, Q2x2+cp Tanta 2, Egypt

REFERENCES:
- [Background] Watchko JF, Tiribelli C. Bilirubin-induced neurologic damage--mechanisms and management approaches. N Engl J Med. 2013 Nov 21;369(21):2021-30. doi: 10.1056/NEJMra1308124. No abstract available. PMID 24256380
- [Background] Usman, F., Diala, U., Shapiro, S., Le Pichon, J.-B., & Slusher, T. Acute bilirubin encephalopathy and its progression to kernicterus: current perspectives. Research and Reports in Neonatology, 8, 33-44 (2018).
- [Background] Watchko JF. Bilirubin-Induced Neurotoxicity in the Preterm Neonate. Clin Perinatol. 2016 Jun;43(2):297-311. doi: 10.1016/j.clp.2016.01.007. Epub 2016 Mar 2. PMID 27235209
- [Background] Das S, van Landeghem FKH. Clinicopathological Spectrum of Bilirubin Encephalopathy/Kernicterus. Diagnostics (Basel). 2019 Feb 28;9(1):24. doi: 10.3390/diagnostics9010024. PMID 30823396
- [Background] Teixeira MH, Borges VMS, Riesgo RDS, Sleifer P. Hyperbilirubinemia impact on newborn hearing: a literature review. Rev Assoc Med Bras (1992). 2020 Jul;66(7):1002-1008. doi: 10.1590/1806-9282.66.7.1002. Epub 2020 Aug 24. PMID 32844928
- [Background] Olds C, Oghalai JS. Audiologic impairment associated with bilirubin-induced neurologic damage. Semin Fetal Neonatal Med. 2015 Feb;20(1):42-46. doi: 10.1016/j.siny.2014.12.006. Epub 2015 Jan 7. PMID 25575899
- [Derived] Zidan LK, Rowisha MA, Nassar MAE, Elshafey RA, El Mahallawi TH, Elmahdy HS. Magnetic resonance spectroscopy and auditory brain-stem response audiometry as predictors of bilirubin-induced neurologic dysfunction in full-term jaundiced neonates. Eur J Pediatr. 2024 Feb;183(2):727-738. doi: 10.1007/s00431-023-05246-z. Epub 2023 Nov 18. PMID 37979048